CLINICAL TRIAL: NCT03241277
Title: Evaluation of Nonsurgical Periodontal Treatment in Patients With Social Phobia: a Randomized Controlled Clinical Trial
Brief Title: Nonsurgical Periodontal Treatment in Patients With Social Phobia
Acronym: NSPTSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33267314.9.0000.0068; 821.780 (Registry Identifier: USaoPauloGH)
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Social Phobia; Periodontal Diseases
Keywords: social phobia; anxiety disorders; DSM-IV TR; periodontal disease; non surgical periodontal treatment
MeSH Terms: conditions — Phobia, Social; Periodontal Diseases; Anxiety Disorders | interventions — Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: Non surgical periodontal treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social phobia (Experimental): Patients with social phobia with no psychiatric treatment Intervention- non surgical periodontal treatment
  Interventions: Procedure: Non surgical periodontal treatment
- Social phobia under Psych T (Experimental): Patients with social phobia under psychiatric treatment (Psych T) Intervention- non surgical periodontal treatment
  Interventions: Procedure: Non surgical periodontal treatment
- Controls (Active Comparator): Patients without social phobia Intervention- non surgical periodontal treatment
  Interventions: Procedure: Non surgical periodontal treatment

INTERVENTIONS:
Procedure: Non surgical periodontal treatment — Scaling and root planning that will be performed with manual curettes or ultrasonic instruments
  Other Names: scaling and root planning

SUMMARY:
Objective: To investigate the impact of nonsurgical periodontal treatment in patients with social anxiety disorder (SAD) and controls without phobia.

DETAILED DESCRIPTION:
Study design: randomized controlled trial. Setting: Institute of Psychiatry from FMUSP (Ipq-FMUSP). Subjects: patients seeking for Social Phobia treatment at IPq-FMUSP ( before and under treatment). Controls: Hospital staff at the HC-FMUSP or volunteers from a list of other studies conducted at the Ipq-FMUSP. Methods: Dental evaluation: probing depth, clinical attachment level and bleeding on probing will be recorded at 6 sites per tooth, as well as the plaque and/or calculus indexes. The number of decayed, missing and filled teeth (DMFT index) will be also assessed. The visual analogue scale (VAS) will be applied for the assessment of pain after probing after the probing recording. Patients will receive a clinical evaluation for halitosis using a Halimeter® to verify the concentration of the volatile sulfur compounds (before and after periodontal treatment). Main psychiatric assessment: Structured Clinical Interview (SCID) for DSM-IV-TR adapted for DSM-5, the Liebowitz Social Anxiety (LSAs). Duration and frequency: after the initial clinical assessment (dental and psychiatric) patients will be randomized into three groups. Two groups (experimental- social phobia with no psychiatric treatment and control) will receive periodontal treatment after the initial psychiatric evaluation. One group will receive periodontal treatment after the improvement of psychiatric condition (3 months after the initial assessment). The non-surgical periodontal treatment will be performed preferably within 24 h. Patients will be reevaluated 3 and 6 months after the end of nonsurgical periodontal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Social Phobia according to the DSM-IV TR adapted for the DSM-5
* Patients with cut-off score of 4 (moderately ill) in the Global Clinical Impression (GCI) rating scale
* Informed consent signature

Exclusion Criteria:

* Patients with severe major depressive disorder at risk for suicide; substance abuse or dependence, psychotic disorders or psychotherapy treatment
* Patients in psychotherapy treatment
* Systemic alteration that precludes periodontal clinical examination

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-10-05 (Estimated); Primary Completion 2019-05-05 (Estimated); Study Completion 2019-10-05 (Estimated)

PRIMARY OUTCOMES:
Probing depth | Change from baseline at 6 months
  the distance from the clinical gingival margin to probe tip

SECONDARY OUTCOMES:
Clinical attachment level | Change from baseline at 6 months
  The distance from cementoenamel junction to probe tip

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Lotufo-Neto, PhD, Study Chair — Faculdade de Medicina FMUSP, Universidade de Sao Paulo, SP, Sao Paulo, SP, BR; Ana Cristina Solis, PhD, Principal Investigator — Faculdade de Medicina FMUSP, Universidade de Sao Paulo, SP, Sao Paulo, SP, BR
Locations (1):
- Department and Institute of Psychiatry - FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Albandar JM, Brunelle JA, Kingman A. Destructive periodontal disease in adults 30 years of age and older in the United States, 1988-1994. J Periodontol. 1999 Jan;70(1):13-29. doi: 10.1902/jop.1999.70.1.13. PMID 10052767
- [Result] Andrade LH, Wang YP, Andreoni S, Silveira CM, Alexandrino-Silva C, Siu ER, Nishimura R, Anthony JC, Gattaz WF, Kessler RC, Viana MC. Mental disorders in megacities: findings from the Sao Paulo megacity mental health survey, Brazil. PLoS One. 2012;7(2):e31879. doi: 10.1371/journal.pone.0031879. Epub 2012 Feb 14. PMID 22348135
- [Result] Armfield JM, Slade GD, Spencer AJ. Dental fear and adult oral health in Australia. Community Dent Oral Epidemiol. 2009 Jun;37(3):220-30. doi: 10.1111/j.1600-0528.2009.00468.x. PMID 19508270
- [Result] Bakri I, Douglas CW, Rawlinson A. The effects of stress on periodontal treatment: a longitudinal investigation using clinical and biological markers. J Clin Periodontol. 2013 Oct;40(10):955-61. doi: 10.1111/jcpe.12142. Epub 2013 Aug 18. PMID 23952266
- [Result] Chung DT, Bogle G, Bernardini M, Stephens D, Riggs ML, Egelberg JH. Pain experienced by patients during periodontal maintenance. J Periodontol. 2003 Sep;74(9):1293-301. doi: 10.1902/jop.2003.74.9.1293. PMID 14584861
- [Result] Claffey N, Polyzois I, Ziaka P. An overview of nonsurgical and surgical therapy. Periodontol 2000. 2004;36:35-44. doi: 10.1111/j.1600-0757.2004.00073.x. No abstract available. PMID 15330942
- [Result] Eke PI, Dye BA, Wei L, Thornton-Evans GO, Genco RJ; CDC Periodontal Disease Surveillance workgroup: James Beck (University of North Carolina, Chapel Hill, USA), Gordon Douglass (Past President, American Academy of Periodontology), Roy Page (University of Washin. Prevalence of periodontitis in adults in the United States: 2009 and 2010. J Dent Res. 2012 Oct;91(10):914-20. doi: 10.1177/0022034512457373. Epub 2012 Aug 30. PMID 22935673
- [Result] Eke PI, Page RC, Wei L, Thornton-Evans G, Genco RJ. Update of the case definitions for population-based surveillance of periodontitis. J Periodontol. 2012 Dec;83(12):1449-54. doi: 10.1902/jop.2012.110664. Epub 2012 Mar 16. PMID 22420873
- [Result] Erovic Ademovski S, Martensson C, Persson GR, Renvert S. The effect of periodontal therapy on intra-oral halitosis: a case series. J Clin Periodontol. 2016 May;43(5):445-452. doi: 10.1111/jcpe.12525. Epub 2016 Apr 18. PMID 26847598
- [Result] Fardal O, Hansen BF. Interviewing self-reported highly anxious patients during periodontal treatment. J Periodontol. 2007 Jun;78(6):1037-42. doi: 10.1902/jop.2007.060407. PMID 17539717
- [Result] Heitz-Mayfield LJ, Lang NP. Surgical and nonsurgical periodontal therapy. Learned and unlearned concepts. Periodontol 2000. 2013 Jun;62(1):218-31. doi: 10.1111/prd.12008. PMID 23574468
- [Result] Khambaty T, Stewart JC. Associations of depressive and anxiety disorders with periodontal disease prevalence in young adults: analysis of 1999-2004 National Health and Nutrition Examination Survey (NHANES) data. Ann Behav Med. 2013 Jun;45(3):393-7. doi: 10.1007/s12160-013-9471-0. PMID 23389686
- [Result] Papapanou PN. The prevalence of periodontitis in the US: forget what you were told. J Dent Res. 2012 Oct;91(10):907-8. doi: 10.1177/0022034512458692. Epub 2012 Aug 30. No abstract available. PMID 22935674
- [Result] Santuchi CC, Cortelli SC, Cortelli JR, Cota LO, Alencar CO, Costa FO. Pre- and post-treatment experiences of fear, anxiety, and pain among chronic periodontitis patients treated by scaling and root planing per quadrant versus one-stage full-mouth disinfection: a 6-month randomized controlled clinical trial. J Clin Periodontol. 2015 Nov;42(11):1024-31. doi: 10.1111/jcpe.12472. Epub 2015 Nov 14. PMID 26461465
- [Result] Sheehan TJ. Creating a psychosocial measurement model from stressful life events. Soc Sci Med. 1996 Jul;43(2):265-71. doi: 10.1016/0277-9536(95)00377-0. PMID 8844930
- [Result] Suhas S, Sudarshan S, Pai KM. "Air bag" organoleptic behavioral experiment for managing fear of oral malodor. J Behav Ther Exp Psychiatry. 2004 Mar;35(1):13-5. doi: 10.1016/j.jbtep.2004.01.001. PMID 15157814
- [Result] Susin C, Valle P, Oppermann RV, Haugejorden O, Albandar JM. Occurrence and risk indicators of increased probing depth in an adult Brazilian population. J Clin Periodontol. 2005 Feb;32(2):123-9. doi: 10.1111/j.1600-051X.2005.00637.x. PMID 15691340
- [Result] Susin C, Haas AN, Oppermann RV, Haugejorden O, Albandar JM. Gingival recession: epidemiology and risk indicators in a representative urban Brazilian population. J Periodontol. 2004 Oct;75(10):1377-86. doi: 10.1902/jop.2004.75.10.1377. PMID 15562916
- [Result] Susin C, Dalla Vecchia CF, Oppermann RV, Haugejorden O, Albandar JM. Periodontal attachment loss in an urban population of Brazilian adults: effect of demographic, behavioral, and environmental risk indicators. J Periodontol. 2004 Jul;75(7):1033-41. doi: 10.1902/jop.2004.75.7.1033. PMID 15341364
- [Result] Vettore M, Quintanilha RS, Monteiro da Silva AM, Lamarca GA, Leao AT. The influence of stress and anxiety on the response of non-surgical periodontal treatment. J Clin Periodontol. 2005 Dec;32(12):1226-35. doi: 10.1111/j.1600-051X.2005.00852.x. PMID 16268999
- [Result] Winkel EG, Roldan S, Van Winkelhoff AJ, Herrera D, Sanz M. Clinical effects of a new mouthrinse containing chlorhexidine, cetylpyridinium chloride and zinc-lactate on oral halitosis. A dual-center, double-blind placebo-controlled study. J Clin Periodontol. 2003 Apr;30(4):300-6. doi: 10.1034/j.1600-051x.2003.00342.x. PMID 12694427
- [Result] de Oliveira Solis AC, Araujo AC, Corchs F, Bernik M, Duran EP, Silva C, Lotufo-Neto F. Impact of post-traumatic stress disorder on oral health. J Affect Disord. 2017 Sep;219:126-132. doi: 10.1016/j.jad.2017.05.033. Epub 2017 May 20. PMID 28549330
- [Result] Liebowitz MR. Social phobia. Mod Probl Pharmacopsychiatry. 1987;22:141-73. doi: 10.1159/000414022. No abstract available. PMID 2885745
- [Result] Lima MS, Soares BG, Paoliello G, Machado Vieira R, Martins CM, Mota Neto JI, Ferrao Y, Schirmer DA, Volpe FM. The Portuguese version of the Clinical Global Impression-Schizophrenia Scale: validation study. Braz J Psychiatry. 2007 Sep;29(3):246-9. doi: 10.1590/s1516-44462007000300010. PMID 17891261